CLINICAL TRIAL: NCT02572843
Title: Anti-PD-L1 Antibody MEDI4736 in Addition to Neoadjuvant Chemotherapy in Patients With Stage IIIA(N2) Non-small Cell Lung Cancer (NSCLC). A Multicenter Single-arm Phase II Trial.
Brief Title: Anti-PD-L1 in Stage IIIA(N2) Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 16/14; 000001480 (Other: SNCTP)
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: NSCLC Non-small Cell Lung Cancer
Keywords: NSCLC; lung cancer; MEDI4736; non-small cell lung cancer; immunotherapy; anti-PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDI4736 (Experimental): Patients whose tumor is deemed resectable at diagnosis will receive 3 cycles (21 days each) of standard chemotherapy with cisplatin/docetaxel followed by 2 cycles (14 days each) of neoadjuvant immunotherapy with MEDI4736 750 mg. Following surgery, patients with complete resection (R0) of their tumor will be administered adjuvant treatment with MEDI4736 750 mg for up to one year or until recurrence, death, unacceptable toxicity or consent withdrawal (whichever occurs first). Patients with incomplete R1/R2 resection, including patients with extracapsular spread of mediastinal lymph node metastases, may undergo standard radiotherapy prior to adjuvant treatment with MEDI4736.
  Interventions: Drug: MEDI4736 (anti-PD-L1)

INTERVENTIONS:
Drug: MEDI4736 (anti-PD-L1) — fixed dosing 750 mg
  Other Names: durvalumab

SUMMARY:
The objective of the trial is to demonstrate that the addition of neoadjuvant and adjuvant immunotherapy (with the anti-PD-L1 antibody MEDI4736) to standard neoadjuvant chemotherapy (with cisplatin/docetaxel) in primary resectable stage IIIA(N2) NSCLC is efficacious and feasible.

DETAILED DESCRIPTION:
Despite multimodal therapy, the cure rate of patients with stage IIIA NSCLC is poor and therapy outcome failed to improve during the past years. The addition of immunotherapy with the anti-PD-L1 antibody MEDI4736 as a novel treatment modality has the potential to improve the outcome without adding substantial toxicity to an otherwise intensive multimodality treatment, as MEDI4736 has been generally well tolerated. Based on the current evidence on immune checkpoint inhibition, there is a strong rationale to test this novel treatment modality also in the curative setting in order to improve local tumor control and prevent distant metastasis to improve the cure rate in this patient population.

The trial investigates the addition of pre- and post-operative immune checkpoint inhibition with MEDI4736 to the previously established standard of care for stage IIIA(N2) patients, which is based on the trials SAKK16/96 and SAKK16/00. Patients whose tumor is deemed resectable at diagnosis will receive 3 cycles (21 days each) of standard chemotherapy with cisplatin (100 mg/m2) / docetaxel (85 mg/m2), followed by 2 cycles (14 days each) of neoadjuvant immunotherapy with MEDI4736 750 mg. Following surgery, patients with complete resection (R0) of their tumor will be administered adjuvant treatment with MEDI4736 750 mg for up to one year or until recurrence, death, unacceptable toxicity or consent withdrawal (whichever occurs first). Patients with incomplete R1/R2 resection, including patients with extracapsular spread of mediastinal lymph node metastases, may undergo standard radiotherapy prior to adjuvant treatment with MEDI4736.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH-GCP regulations before patient registration and any protocol-related procedures.
* Pathologically proven NSCLC (adeno-, squamous-, large cell carcinoma or NSCLC not otherwise specified) irrespective of genomic aberrations or PD-L1 expression status.
* Tumor tissue is available for the mandatory translational research (preferably histology, cytology allowed).
* Tumor stage T1-3N2M0 (stage IIIA(N2)) according to the TNM classification, 7th edition, (October 2009). Mediastinal lymph node staging has to follow the process chart.
* Tumor is considered resectable based on a multidisciplinary tumor board decision made before neoadjuvant treatment. Resectable is when a complete resection can be achieved according to Rami-Porta {Rami-Porta, 2005 #88}.
* Measurable disease according to RECIST 1.1 criteria (non-nodal lesions ≥10 mm in longest diameter, lymph nodes ≥15 mm in short axis) by PET/CT with contrast enhanced CT-scan.
* WHO performance status 0-1.
* Age 18-75 years at time of registration.
* Appropriate lung function based on the ESTS guidelines {Brunelli, 2009 #19}:

  * For pneumonectomy: FEV1 and DLCO ≥80%. If one of both <80% an exercise test peak VO2 >75% or 20ml/kg/min is needed,
  * For resection less than pneumonectomy (resection up to the calculated extent): exercise test peak VO2 ≥35% or ≥10ml/kg/min, with predicted postoperative FEV1 and DLCO ≥ 30%.
* Adequate hematological values: hemoglobin ≥ 90 g/L, absolute neutrophils count ≥ 1.5 x 109/L, platelets count ≥ 100 x 109/L.
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 1.5 x ULN, AP ≤ 2.5 x ULN.
* Adequate renal function: calculated creatinine clearance ≥ 60 mL/min, according to the formula of Cockcroft-Gault.
* Women with child-bearing potential are using effective contraception are not pregnant or lactating and agree not to become pregnant during participation in the trial and during 90 days after the last treatment. A negative serum pregnancy test performed within 7 days before registration into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and during 90 days after the last treatment.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

* Presence of any distant metastasis or N3 disease. Brain metastases have to be excluded by CT or MRI.
* Sulcus superior tumors (Pancoast tumors).
* Previous or concomitant malignancy within 5 years prior registration with the exception of adequately treated localized non-melanoma skin cancer or cervical carcinoma in situ.
* Any previous treatment for NSCLC.
* Any previous treatment with a PD-1 or PD-L1 inhibitor, including MEDI4736.
* Previous radiotherapy to the chest.
* Absolute contraindications for the use of corticosteroids as premedication.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to registration.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (i.e. which must not exceed 10 mg/day of prednisone or an equivalent corticosteroid) and the premedication for chemotherapy.
* Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 3 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's Correction.
* Preexisting peripheral neuropathy (> grade 1).
* Body weight less than 30 kg.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: - Vitiligo or resolved childhood asthma/atopy - Hypothyroidism stable on hormone replacement or Sjorgen's syndrome
* Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis).
* Known evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* Known history of previous clinical diagnosis of tuberculosis.
* Receipt of live attenuated vaccination any time during trial therapy with MEDI4736 and within 30 days of receiving the last dose of MEDI4736.
* Any concomitant drugs contraindicated for use with MEDI4736: this includes systemic corticosteroids, methotrexate, azathioprine, and tumor necrosis factor (TNF)-α blockers. Any concomitant drugs contraindicated for use with the other trial drugs according to the locally approved product information.
* Known hypersensitivity to trial drugs (cisplatin and docetaxel), to the IMP or to any excipient.
* Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, severe hearing impairment), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sacha Rothschild, MD, PhD, Study Chair — University Hospital, Basel, Switzerland
Locations (19):
- Switzerland (19):
  - Stadtspital Triemli, Zurich, Canton of Zurich
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - St. Claraspital Basel, Basel
  - Universitaetsspital Basel, Basel
  - IOSI Ospedale Regionale di Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Spital Thurgau AG, Frauenfeld
  - Hopital Fribourgeois HFR, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - CCAC Lausanne, Lausanne
  - Centre hospitalier universitaire vaudois CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden Onkozentrum Zürich, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmid D, Sobottka B, Manzo M, Trub M, Leonards K, Herzig P, Oyewole OR, Jermann P, Hayoz S, Savic Prince S, Tochtermann G, Natoli M, Pless M, Bettini A, Fruh M, Mauti LA, Britschgi C, Peters S, Mark M, Ochsenbein AF, Janthur WD, Waibel C, Mach N, Froesch P, Buess M, Bohanes P, Gonzalez M, Alborelli I, Rothschild SI, Koelzer VH, Zippelius A. Tumor immune dynamics and long-term clinical outcome of stage IIIA NSCLC patients treated with neoadjuvant chemoimmunotherapy. Nat Commun. 2025 Sep 30;16(1):8673. doi: 10.1038/s41467-025-63696-5. PMID 41027867
- [Derived] Rothschild SI, Zippelius A, Eboulet EI, Savic Prince S, Betticher D, Bettini A, Fruh M, Joerger M, Lardinois D, Gelpke H, Mauti LA, Britschgi C, Weder W, Peters S, Mark M, Cathomas R, Ochsenbein AF, Janthur WD, Waibel C, Mach N, Froesch P, Buess M, Bohanes P, Godar G, Rusterholz C, Gonzalez M, Pless M; Swiss Group for Clinical Cancer Research (SAKK). SAKK 16/14: Durvalumab in Addition to Neoadjuvant Chemotherapy in Patients With Stage IIIA(N2) Non-Small-Cell Lung Cancer-A Multicenter Single-Arm Phase II Trial. J Clin Oncol. 2021 Sep 10;39(26):2872-2880. doi: 10.1200/JCO.21.00276. Epub 2021 Jul 12. PMID 34251873

RESULTS

PARTICIPANT FLOW:
Period: Accrual
Arm/Group | MEDI4736
Started | 68
Completed | 67
Not Completed | 1
Not completed — Brain metastasis retrospectively detected | 1
Period: Neoadjuvant chemotherapy
Arm/Group | MEDI4736
Started | 67
Completed | 62
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Starting subsequent treatment due progressive disease clinically assessed | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 1
Period: Neoadjuvant immunotherapy
Arm/Group | MEDI4736
Started | 62
Completed | 58
Not Completed | 4
Not completed — Progressive disease | 2
Not completed — Withdrawal by Subject | 1
Not completed — General status and respiratory capacity diminution | 1
Period: Surgery
Arm/Group | MEDI4736
Started | 58
Completed | 50
Not Completed | 8
Not completed — lost to follow up | 7
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: FAS
Arm/Group | MEDI4736
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 67

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Rate
Description: Measured using the Kaplan-Meier method
Time Frame: at 12 months
Population: FAS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 67
percentage of participants | 73.4 [62.7 to 81.5]

2. Secondary Outcome: Median Event-free Survival (EFS)
Description: Measured using the Kaplan-Meier method
Time Frame: up to 7 years from registration
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | MEDI4736
Number analyzed (Participants) | 67
years | 4.0 [2.4 to NA] — Not reached due to insufficient number of participants with events

3. Secondary Outcome: Overall Survival (OS) Rate
Description: Measured using the Kaplan-Meier method
Time Frame: at 1, 2, 3, 4 & 5 years after registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 67
percentage of participants
  OS rate at 1 year | 91.0 [81.0 to 95.8]
  OS rate at 2 years | 83.3 [71.8 to 90.4]
  OS rate at 3 years | 70.7 [58.0 to 80.2]
  OS rate at 4 years | 67.5 [54.6 to 77.5]
  OS rate at 5 years | 65.8 [52.9 to 76.0]

4. Secondary Outcome: Objective Response (OR) After Neoadjuvant Chemotherapy (FAS)
Time Frame: After Neoadjuvant Chemotherapy, up to 3 months
Population: patients who received neoadjuvant chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 67
percentage of participants | 43.3 [31.2 to 56.0]

5. Secondary Outcome: Objective Response (OR) After Neoadjuvant Immunotherapy (FAS II)
Description: Measured using the Kaplan-Meier method
Time Frame: After Neoadjuvant immunotherapy, up to 3 months
Population: patients who received neoadjuvant immunotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 62
percentage of participants | 58.1 [44.8 to 70.5]

6. Secondary Outcome: Pathological Responses (pCR)
Time Frame: at 12 months
Population: the 55 resected patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MEDI4736
Number analyzed (Participants) | 55
percentage of participants | 18.2 [9.1 to 30.9]

7. Secondary Outcome: Adverse Events (AEs) (According to NCI CTCAE v4.0)
Description: Outcomes are described under "Adverse events".
Time Frame: Adverse events were recorded from registration up to 13 months after surgery, up to 17 months. Deaths were reported up to 8 years from registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from registration up to 13 months after surgery, up to 17 months. Deaths were reported up to 8 years from registration
Arm/Group | MEDI4736
All-Cause Mortality (participants affected / at risk) | 25/67
Serious Adverse Events (participants affected / at risk) | 36/67
Other Adverse Events (participants affected / at risk) | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 (N=67)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pseudomembranous colitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infection of unknown origin (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 6 (7)
Mucosal infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury to superior vena cava (Injury, poisoning and procedural complications) | 1 (1)
Postoperative pulmonary leak and lung infection (Injury, poisoning and procedural complications) | 1 (1)
Alt increased, ast increased, ggt increased (Injury, poisoning and procedural complications) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nsclc (adenocarcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenopathy surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 (N=67)
Anemia (Blood and lymphatic system disorders) | 7 (12)
Hearing impaired (Adults) (Ear and labyrinth disorders) | 7 (8)
Tinnitus (Ear and labyrinth disorders) | 24 (26)
Vertigo (Ear and labyrinth disorders) | 6 (6)
Hyperthyroidism (Endocrine disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 4 (5)
Conjunctivitis (Eye disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 16 (23)
Constipation (Gastrointestinal disorders) | 25 (38)
Diarrhea (Gastrointestinal disorders) | 42 (71)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 (10)
Mucositis oral (Gastrointestinal disorders) | 8 (12)
Nausea (Gastrointestinal disorders) | 45 (80)
Stomach pain (Gastrointestinal disorders) | 6 (11)
Vomiting (Gastrointestinal disorders) | 29 (47)
Chills (General disorders) | 6 (7)
Edema limbs (General disorders) | 9 (12)
Fatigue (General disorders) | 46 (77)
Fever (General disorders) | 9 (12)
Flu like symptoms (General disorders) | 7 (9)
Non-cardiac chest pain (General disorders) | 11 (13)
Pain (General disorders) | 24 (39)
Bronchial infection (Infections and infestations) | 5 (5)
Lung infection (Infections and infestations) | 8 (10)
Mucosal infection (Infections and infestations) | 6 (8)
Rhinitis infective (Infections and infestations) | 4 (4)
Upper respiratory infection (Infections and infestations) | 5 (7)
Urinary tract infection (Infections and infestations) | 8 (16)
Creatinine increased (Investigations) | 7 (12)
Neutrophil count decreased (Investigations) | 7 (11)
Platelet count decreased (Investigations) | 6 (9)
White blood cell decreased (Investigations) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 27 (43)
Hyponatremia (Metabolism and nutrition disorders) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Dizziness (Nervous system disorders) | 6 (7)
Dysesthesia (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 36 (50)
Headache (Musculoskeletal and connective tissue disorders) | 12 (17)
Paresthesia (Nervous system disorders) | 8 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (27)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 17 (19)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (46)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (44)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 36 (39)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (18)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (10)
Hypertension (Vascular disorders) | 7 (13)
Hypotension (Vascular disorders) | 4 (5)
Thromboembolic event (Vascular disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02572843/Prot_SAP_000.pdf